CLINICAL TRIAL: NCT04681196
Title: Evaluation of Different Effects of Nasal Versus Oronasal Mask in Continuous Positive Airway Pressure (CPAP) Treatment of Patients Affected by Obstructive Sleep Apnea Syndrome (OSAS).
Brief Title: Nasal Versus Oronasal Mask in Continuous Positive Airway Pressure (CPAP) Treatment of Patients Affected by Obstructive Sleep Apnea Syndrome (OSAS).
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Francesco Tavalazzi, Francesco Tavalazzi Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 195/2020/Oss/AOUBO
Record Dates: First submitted 2020-11-20; First posted 2020-12-23 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Osa Syndrome
Keywords: OSAS; CPAP; nasal mask; oronasal mask
MeSH Terms: conditions — Carnevale syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients affected by OSA treated with CPAP / paradox effect group: patients with obstructive sleep apnea, exhibiting persistent obstructive events and paradoxical obstruction when wearing oronasal masks during CPAP, that were fully recovered with the shift to nasal one with the same or also lower pressure
  Interventions: Other: patients shifted to nasal mask after persistent OSA with oronasal mask
- patients affected by OSA treated with CPAP / control group (no paradox effect): patients with obstructive sleep apnea, with no obstructive events when wearing oronasal masks during CPAP

INTERVENTIONS:
Other: patients shifted to nasal mask after persistent OSA with oronasal mask — In this group were selected OSA patients exhibiting persistent obstructive events and paradoxical obstruction with oronasal masks during CPAP , that were fully recovered (no more OSA detected) with the shift to nasal one
  Groups: patients affected by OSA treated with CPAP / paradox effect group

SUMMARY:
Continuous positive airway pressure (CPAP) is considered the gold standard treatment for patients with moderate to severe obstructive sleep apnea (OSA).

Nasal and oronasal masks are often used interchangeably and are generally believed to be equally effective; the choice of interface for OSA therapy remains largely based on clinical judgement and patients preference. However, there is increasing evidence that CPAP delivered by an oronasal mask may be less effective, requires more pressure and are worse tolerated than nasal mask. Patients with OSA on oronasal mask are also less adherent to CPAP.

Some authors have suggested that in some subjects, the CPAP was not effective when an oronasal mask was used. Moreover when pressures are increased to overcome the obstruction, a paradoxical obstruction may take place.

Specific mechanisms explaining upper-airway obstruction events remain unclear and it is not known how many patients exhibit this behavior.

This observational retrospective study is designed to compare a group of patients with obstructive sleep apnea with persistent obstructive events using oronasal masks during CPAP, that were fully recovered with the shift to nasal one with the same or also lower pressure, versus a control group of patients who did not report obstruction with oronasal masks. Aim of the study was to find differences in term of clinical, anatomical and physiological characteristics between these two groups.

DETAILED DESCRIPTION:
Continuous positive airway pressure (CPAP) is considered the gold standard treatment for patients with moderate to severe obstructive sleep apnea (OSA).

The treatment of OSA with CPAP was first proposed by Sullivan et al and traditionally delivered using a nasal mask because the pressure applied through the nose would be transmitted as a pneumatic splint to the back of the upper airway and would push them anteriorly.

However patients with OSA frequently present nasal obstruction and leakage of air from the mouth, and different mask interfaces have been developed, including the oronasal mask that may be used to deliver CPAP.

Nasal and oronasal masks are often used interchangeably and are generally believed to be equally effective; the choice of interface for OSA therapy remains largely based on clinical judgement and patients preference .

In our clinical practice, CPAP titration is started adapting the patient to a nasal mask but an oronasal can be selected if a patient reports inability to breathe through their nose, severe nasal obstruction, leakage of air from the mouth or from other part of the face due to anatomical variation.

However, there is increasing evidence that CPAP delivered by an oronasal mask may be less effective, requires more pressure and are worse tolerated than nasal mask.

Patients with OSA on oronasal mask are also less adherent to CPAP. One recent randomised trial and a preliminary report suggest that subjects with sleep apnea treated with CPAP showed a significantly lower residual AHI when subjects wore a nasal mask rather than a oronasal mask.

Similarly, a recent prospective observational cohort study suggested that the use of a facial mask was associated with higher CPAP pressure requirements than both nasal masks and nasal pillows.

Some authors have suggested that in some subjects, the CPAP was not effective when an oronasal mask was used. Moreover when pressures are increased to overcome the obstruction, a paradoxical obstruction may take place.

These findings have been called "the Starling paradox effect", according to which the pressure that opens the pharynx can also lead to pharyngeal collapse when applied orally.

In these difficult-to-titrate patients the specific mechanisms explaining upper-airway obstruction events remain unclear and it is not known how many patients exhibit this behavior.

This observational retrospective study is designed to compare a group of patients with obstructive sleep apnea with persistent obstructive events using oronasal masks during CPAP, that were fully recovered with the shift to nasal one with the same or also lower pressure, versus a control group of patients who did not report obstruction with oronasal masks.

Aim of the study was to find differences in term of clinical, anatomical and physiological characteristics between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of OSA and use of CPAP treatment
* age> or equal to 18 years old
* sign of informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this observational retrospetive study were selected patients affected by OSA treated with CPAP. From this population were selected patients using oronasal mask with complete recovery of OSA (AHI<5) during CPAP treatment (control group) and patients shifted to nasal mask due to persistent of obstructive events (AHI>5) during the initial treatment with oronasal mask.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
differences in terms of age between groups | Up to one month.
  differences in terms of age (measured in years) between patients with paradox effect versus patients without paradox effect (control group); age considered at the time of OSA diagnosis
differences in terms of body mass index between groups | Up to one month.
  differences in terms of body mass index (BMI), measured in Kg/m2, between patients with paradox effect versus patients without paradox effect (control group); BMI considered at the time of OSA diagnosis.
differences in terms of basal value of apnea-hypopnea index (OSA severity) between groups | Up to one month.
  differences in terms of basal value of apnea-hypopnea index (OSA severity) between groups. AHI considered at the time of OSA diagnosis (basal cardio-respiratory monitoring) Apnea-hypopnea index (AHI) measures number of obstructive events (apnea and hypopnea) per hour during basal cardio-respiratory monitoring. AHI> 5 is diagnostic of OSA. Severity of OSA is proportional to AHI value.
differences in terms of basal value of minimum and mean nocturnal oxygen saturation between groups. | Up to one month.
  differences in terms of basal value of minimum and mean nocturnal oxygen saturation (respectively minimum SpO2 % and mean SpO2 %) between groups.Minimum and mean Oxygen Saturation considered at the time of OSA diagnosis (basal cardio-respiratory monitoring).
differences in terms of basal value of time spent under SpO2<90% and under SpO2<80% between groups. | Up to one month.
  differences in terms of basal value of time spent under SpO2<90% (CT90) and under SpO2<80% (CT80) between groups.minimum and mean Oxygen Saturation considered at the time of OSA diagnosis (basal cardio-respiratory monitoring).
  These two parameters are expressed as % of total registration time during basal cardio-respiratory monitoring at the time od OSA diagnosis.
differences in terms of oxygen desaturation index between groups. | Up to one month.
  differences in terms of oxygen desaturation index (ODI) between groups. ODI represents number of decline of SpO2 > or equal to 3% events per hours during basal cardio-respiratory monitoring collected at the time od OSA diagnosis.ODI considered at the time of OSA diagnosis (basal cardio-respiratory monitoring)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico S. Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No